CLINICAL TRIAL: NCT01724814
Title: A First-in-human Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of HM12460A
Acronym: HM12460A
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HM-INS-101
Record Dates: First submitted 2012-11-05; First posted 2012-11-12 (Estimated); Last update posted 2017-11-08 (Actual); Status verified 2017-11

CONDITIONS: Healthy; Type 1 Diabetes Mellitus; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Cohort S1 (Experimental): HM12460A Dose 1 (1.2 nmol/kg) or placebo
  Interventions: Drug: HM12460A; Drug: Placebo
- Cohort S2 (Experimental): HM12460A Dose 2 (2.4 nmol/kg) or Placebo
  Interventions: Drug: HM12460A; Drug: Placebo
- Cohort S3 (Experimental): HM12460A Dose 3 (4.8 nmol/kg) or Placebo
  Interventions: Drug: HM12460A; Drug: Placebo
- Cohort S4 (Experimental): HM12460A Dose 4 (9.6 nmol/kg) or Placebo
  Interventions: Drug: HM12460A; Drug: Placebo
- Cohort S5 (Experimental): HM12460A Dose 5 (14.4 nmol/kg) or Placebo
  Interventions: Drug: HM12460A; Drug: Placebo
- Cohort S6 (Experimental): HM12460A Dose 6 (19.2 nmol/kg) or Placebo
  Interventions: Drug: HM12460A; Drug: Placebo

INTERVENTIONS:
Drug: HM12460A — Single dose SC administration ranging from 1.2 nmol/kg to 19.2 nmol/kg of HM12460A
  Other Names: LAPS-Insulin
Drug: Placebo — Singe dose SC administration of Placebo

SUMMARY:
Study Design:

Part 1.Randomized, double-blind, placebo-controlled, escalating single-dose design with Healthy volunteers Part 2.Open , sequential, two-period, single dose study with type 1 diabetes Part 3.Open, sequential, two-period, single dose study with type 2 diabetes

DETAILED DESCRIPTION:
The principle objectives of this study are to assess safety and tolerability and to explore pharmacokinetic(PK) and pharmacodynamic(PD) parameters of a single dose of a novel very-long acting insulin formulation (HM12460A) in comparison to a single dose of human Neutral Protamine Hagedorn (NPH) in healthy volunteers (part 1), subjects with type 1 diabetes (part 2) and in subjects with type 2 diabetes (part 3).

The study will incorporate adaptive elements to provide both PK and PD data. The dose of HM12460A to be administered to the subjects with type 1 diabetes and type 2 diabetes will be guided by PK data from part 1 of the study; the PD assessment of HM12460A in subjects with diabetes will also be informed by knowledge of PK gained from the healthy volunteer study.

ELIGIBILITY:
Inclusion Criteria:

Healthy subjects

* Age ≥18 and ≤70 years
* Non-obese; body mass index between 18.0 and 30.0 kg/m2 inclusive.
* Considered generally healthy upon completion of medical history, physical examination and biochemical investigations as judged by the Investigator.
* Non-smoker, or light smoker, defined as <15 cigarettes/day and able to abstain from smoking during confinement period.
* Females must be non-pregnant and non-lactating, and either surgically sterile (e.g., tubal occlusion, hysterectomy, bilateral salpingectomy, bilateral oophorectomy) or post-menopausal for >12 months. Males must be surgically sterile, abstinent or if engaged in sexual relations of child-bearing potential, the subject must be using an acceptable contraceptive method during and for during a period of 60 days after the last dose of Study Drug.
* Signed and dated informed consent obtained before any trial-related activities. (Trial-related activities are any procedure that would not have been performed during normal management of the subject).

Exclusion Criteria:

* Previous participation in this trial or other clinical trials within the last 3 months.
* Clinically significant abnormal hematology or biochemistry screening tests, as judged by the Investigator. In particular, healthy subjects with liver enzymes above the upper limit of the normal range and subjects with diabetes who have elevated liver enzymes (AST or ALT >2 times the upper limit of normal) or impaired renal function (elevated serum creatinine values above the upper limit of normal) will be excluded.
* History of any illness that, in the opinion of the Investigator, might confound the results of the trial or pose risk in administering the trial drug to the subject. In particular, subjects with significant cardiovascular disease, anemia (hemoglobin below the lower limit of normal) or hemoglobinopathy will not be allowed to enter the trial.
* Clinically significant abnormal ECG at screening, as judged by the Investigator.
* History of alcohol abuse.
* Any positive reaction of drugs of abuse.
* Hepatitis B or C or HIV positive.
* Use of prescription drugs within 3 weeks preceding the first dosing of insulin, except for medications deemed acceptable per protocol specific list of concomitant medications.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2012-12-20 (Actual); Primary Completion 2014-07-01 (Actual); Study Completion 2014-07-01 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of treatment emergent adverse events | one year

SECONDARY OUTCOMES:
Peak Plasma Concentration(Cmax) of HM12460A following a single dose in Parts 1-3 | one year
  PK properties of HM12460A following a single dose in Parts 1-3 will be assessed in plasma using a validated assay

CONTACTS AND LOCATIONS:
Locations (1):
- Hanmi pharma, Chula Vista, California, United States